CLINICAL TRIAL: NCT07105813
Title: A Clinical Trial of the Safety and Efficacy of a Perforated Surgical Navigation and Localization System for Use in Percutaneous Pulmonary Ablation of Multiple Ground-glass Nodules
Brief Title: A Clinical Trial of Percutaneous Lung Ablation Using Navigational Positioning Robot-assisted Procedures
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Xiaolong Yan, Dr. (Other)
Responsible Party: Sponsor-Investigator, Xiaolong Yan, Dr., Deputy Chief Physician, Department of Thoracic Surgery, Tangdu Hospital, Air Force Military Medical University. PhD, Researcher, Doctoral and Postdoctoral Supervisor, Deputy Chief of Thoracic Surgery, Tangdu Hospital, Tang-Du Hospital
Organization: Tang-Du Hospital (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: WD-2024SY-1001
Record Dates: First submitted 2025-07-09; First posted 2025-08-06 (Actual); Last update posted 2025-08-06 (Actual); Status verified 2025-07

CONDITIONS: Percutaneous Lung Ablation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Navigational Positioning System for Puncture Surgery (Experimental)
  Interventions: Device: Navigational Positioning System for Puncture Surgery

INTERVENTIONS:
Device: Navigational Positioning System for Puncture Surgery — Suitable for puncture surgery navigation and localization systems to assist in the procedure

SUMMARY:
The purpose of the trial is to exploratively evaluate the safety and efficacy of the Puncture Surgery Navigation and Positioning System for CT-guided percutaneous lung ablation procedures for multiple ground glass nodules.

Thirty subjects are planned to be enrolled in this study. In the study, it is planned to perform CT-guided percutaneous lung ablation procedures in the enrolled patients using the Puncture Surgery Navigation and Positioning System, and to evaluate the technical success rate, puncture accuracy, one-time technical success rate, one-needle penetration in place, number of needle adjustments, time to puncture, and complication rate

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥18 years and <80 years, regardless of sex;
2. Diagnosis of persistent multiple pulmonary ground glass nodules (GGN), including pure ground glass nodules (pGGN) and mixed ground glass nodules (mGGN), with no limitation on the size and number of nodules, where persistence is defined as the non-resolution of the GGN after 3 months of follow-up after detection;
3. Patients who are evaluated as needing treatment for a primary or secondary lesion of a ground glass nodule in the lung, and the diameter of the lesion to be ablated is ≥6.0 mm, and who meet any of the following can be enrolled:

   1. Cannot tolerate surgical resection due to poor cardiopulmonary function or advanced age;
   2. Refuse to undergo surgical resection;
   3. Residual lesions or new lesions after surgical resection;
   4. Severe pleural adhesions or pleural cavity atresia from various causes;
   5. Single lung (absence of one side of the lung from various causes);
   6. Severe anxiety that is not relieved by psychological or pharmacological treatment.
4. The patient fully understands the benefits and risks of this trial, is willing to participate in the trial and signs an informed consent form.

Exclusion Criteria:

1. Those with skin redness, swelling, broken skin, symptoms of skin diseases at the puncture site, dermatologic diseases that cannot be affixed with markers, or acute suppurative infections in the pleural cavity;
2. Platelets <50 × 109/L, or severe bleeding tendency, coagulation dysfunction that cannot be corrected in a short period of time (prothrombin time >18 s, plasminogen activity <40%), or anticoagulant therapy and/or antiplatelet drugs that have not been discontinued for more than 5 d to 7 d prior to ablation, and the interval between the last use of bevacizumab has not exceeded 1 month;
3. Those with severe systemic infection and high fever (>38.5°C);
4. Lung nodules close to important organs such as mediastinum or cardiac great vessels;
5. Those who have other diseases such as pulmonary pustules or pulmonary cysts leading to pneumothorax in the proposed puncture path, or those who have obvious infectious lesions in the puncture path;
6. Those with poorly controlled pleural effusion;
7. Severe pulmonary fibrosis and pulmonary hypertension;
8. Those with severe cardiac, hepatic, pulmonary, renal, or cerebral insufficiency;
9. Those with severe anemia, dehydration, and severe disorders of nutritional metabolism that cannot be corrected or improved in the short term;
10. Those with an Eastern Cooperative Oncology Group (ECOG) score >3;
11. Patients with episodic psychosis;
12. Those with a combination of other tumors with extensive metastases and an expected survival of <6 months;
13. Those who cannot cooperate, those who cannot control cough, and those who cannot tolerate puncture;
14. Women who are in pregnancy or breastfeeding, and others who cannot receive intraoperative radiation;
15. Those who have participated or are participating in another clinical trial within 28 days prior to screening;
16. Subjects who are assessed by the investigator to have poor compliance or other reasons why they should not participate in the trial.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 30 (Estimated)
Dates: Start 2025-09-15 (Estimated); Primary Completion 2026-12-30 (Estimated); Study Completion 2026-12-30 (Estimated)

PRIMARY OUTCOMES:
Technical success rate | Perioperative/Periprocedural
  Researchers successfully completed percutaneous ablation surgery using a robotic system. If there were no major needle adjustments during the procedure and no instrument defects or mechanical arm collisions occurred, the technique can be deemed successful.

SECONDARY OUTCOMES:
The proportion of cases where puncture is successful after one puncture or fine adjustment | Perioperative/Periprocedural
One technical success rate | Perioperative/Periprocedural
  A technical success is defined as the achievement of technical success with a single needle puncture or minor adjustments. One technical success rate is the percentage of technical success cases in the total number of cases.
One-needle puncture placement rate | Perioperative/Periprocedural
  After the needle is inserted according to the pre-planned puncture direction, angle, and depth, a CT scan is performed to observe the positional relationship between the needle tip and the lung nodule. If the proposed ablation range at the needle tip position can surround the lung nodule by 5-10 mm, the researcher determines that no needle adjustment is necessary and that the ablation procedure can continue, thus confirming that the needle is in the correct position. The one-needle puncture success rate is the proportion of punctures that are successful on the first attempt.
Complete ablation rate | Perioperative/Periprocedural
  By measuring whether the post-ablation GGO exceeds the pre-ablation GTR boundary by 5-10 mm on the post-ablation CT image, it is determined whether complete ablation has been achieved.
Number of needle adjustments | Perioperative/Periprocedural
puncture duration | Perioperative/Periprocedural
Adverse event rate | Perioperative/Periprocedural
Incidence of device defects | Perioperative/Periprocedural